CLINICAL TRIAL: NCT06262698
Title: The Effect of Simulation-Based Education on Nursing StudentsCAM Knowledge, Attitudes, and Health Beliefs Regarding Medication Use: A Randomized Controlled Study
Brief Title: The Effect of HBM-Based Education on Nursing Students
Acronym: HBM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Gönül GÖKÇAY, Asist. Prof., Kafkas University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 81825902.903/148
Record Dates: First submitted 2024-02-06; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Nursing; Evidence-Based Nursing
Keywords: Nursing student; Health Belief Model; Traditional and Complementary Medicine; knowledge; attitudes; Health belief related to medication use; complementary and alternative medicine
MeSH Terms: conditions — Behavior | interventions — Evaluation Studies as Topic

STUDY DESIGN:
Intervention Model Description: The experimental group will receive six weeks of HBM-based training.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants were assigned to groups using the "simple randomization method". Participants were not informed of which group they were in. Automated computer-based randomization resulted in the implementation of the experiment with the scheduling scenario and confidential allocation of participants to one of the four intervention branches. The researcher was blind to all conditions until the participants started the computer program and the intervention began. Participants were also unaware of whether the group they were assigned to was an experimental or a control condition. In addition, researchers coding and analyzing data will be blind to randomization and interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): "Based on the SIM model, the intervention group will receive 6 sessions of training (each session lasting 40 minutes). The training sessions will be as follows:
  1. st Session: Traditional/Alternative medical systems
  2. nd Session: Mental-physical interventions
  3. rd Session: Biologically based treatments
  4. th Session: Manipulative and physical-based therapies
  5. th Session: Energy therapies
  6. th Session: Training on proper prescription drug use"
  Interventions: Behavioral: Experiment group; Other: Pre-post test
- Control (Other): Nursing students will receive their regular semester courses; no additional intervention will be implemented.
  Interventions: Other: Pre-post test

INTERVENTIONS:
Behavioral: Experiment group — The experimental group will receive six weeks of HBM-based training.
  Arms: experimental
Other: Pre-post test — The TCM Attitude Scale (CACMAS), Medication Health Belief Scale

SUMMARY:
The purpose of the study is to investigate the effect of HBM-based education on CAM knowledge, attitudes, and health beliefs related to medication use among nursing students through a randomized controlled trial.

Research hypotheses:

Hypothesis 01: There is no effect of HBM-based education on CAM knowledge level among nursing students.

Hypothesis 1: There is an effect of HBM-based education on CAM knowledge level among nursing students.

Hypothesis 02: There is no effect of HBM-based education on CAM attitude level among nursing students.

Hypothesis 2: There is an effect of HBM-based education on CAM attitude level among nursing students.

Hypothesis 03: There is no effect of HBM-based education on health beliefs related to medication use among nursing students.

Hypothesis 3: There is an effect of HBM-based education on health beliefs related to medication use among nursing students.

DETAILED DESCRIPTION:
The Complementary and Alternative Medicine (CAM), according to the World Health Organization, encompasses knowledge, skills, and practices based on the beliefs and experiences of different cultures for the prevention, diagnosis, treatment, and preservation of health for physical and mental ailments. Reasons for the use of CAM today include its perceived assistance in chronic, psychiatric, and end-stage diseases where conventional medicine may not provide a complete solution, patients' desire for control over their treatments, cultural compatibility and accessibility, and the simplicity of procedures, often with minimal or no invasiveness.The aim of this project is to determine the impact of HBM-based education provided to nursing students on their knowledge, attitude, and health beliefs related to CAM and medication use through a randomized controlled study. It is planned to be conducted between January 2024 and December 2024. The project will involve a total of 120 students in intervention and control groups. Data collection instruments will include a pre-test Personal Information Form, CAM Knowledge and Attitude Scale, Medication Beliefs Scale, and post-test CAM Knowledge and Attitude Scale, Medication Beliefs Scale after six weeks of education.Through this project, the importance of CAM practices for healthcare professionals, especially nursing candidates, will be emphasized. The study will explore various application areas of CAM based on cultural and belief contexts by examining commonly used CAM methods for disease treatment and health preservation. This study will serve as an important resource for assessing the knowledge and attitudes of healthcare professionals, particularly nursing candidates, regarding CAM, understanding the use of complementary practices in healthcare, and raising awareness among healthcare professionals.The popularity of CAM practices, patients' interest in complementary treatments, and the role of these treatments in healthcare underscore the importance of including CAM education in nursing curricula. Additionally, the research will demonstrate how CAM can be evaluated using the Health Belief Model (HBM) and how nursing candidates' knowledge, attitudes, and beliefs toward such practices are shaped. The results of the study may contribute significantly to evaluating the effectiveness of educational programs designed to increase nursing candidates' knowledge levels and influence their attitudes toward CAM.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the nursing program at Kafkas University
* Willing to participate in the study voluntarily

Exclusion Criteria:

* - Choosing not to participate in the study voluntarily

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The TCM Attitude Scale (CACMAS) The GETAT Attitude Scale (CACMAS): The scale, developed by McFadden et al. (2010), consists of 27 items rated on a 7-point Likert scale. Its Turkish validity and reliability were established by Köse et al. (2018). | three months
  The scale, developed by McFadden et al. (2010), consists of 27 items rated on a 7-point Likert scale. Its Turkish validity and reliability were established by Köse et al. (2018).The high score on the scale indicates a high level of knowledge and attitude towards TCM.
The Medication Health Belief Scale | three months
  Validity and reliability of the scale were established by Erci and Çiçek (2012). The scale consists of 35 items and comprises 6 sub-dimensions. The minimum score that can be obtained from the scale is 35, and the maximum score is 175. The high score on the scale indicates a strong belief in health regarding prescription drug use.

CONTACTS AND LOCATIONS:
Overall Officials: Gönül GÖKÇAY, Asist. Prof., Principal Investigator — Kafkas University-Kafkas University Faculty of Health Sciences; İlknur ÇİÇEK, Student, Study Chair — Kafkas University-Kafkas University Faculty of Health Sciences
Locations (1):
- Kafkas University Faculty of Health Sciences, Kars, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kemppainen LM, Kemppainen TT, Reippainen JA, Salmenniemi ST, Vuolanto PH. Use of complementary and alternative medicine in Europe: Health-related and sociodemographic determinants. Scand J Public Health. 2018 Jun;46(4):448-455. doi: 10.1177/1403494817733869. Epub 2017 Oct 4. PMID 28975853
- [Result] Bodeker G, Kronenberg F. A public health agenda for traditional, complementary, and alternative medicine. Am J Public Health. 2002 Oct;92(10):1582-91. doi: 10.2105/ajph.92.10.1582. PMID 12356597